CLINICAL TRIAL: NCT04961710
Title: Extension Study of Hetrombopag Olamine in Patients With Treatment-naive Severe Aplastic Anemia
Brief Title: Extension Study of Hetrombopag in Severe Aplastic Anemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-TPO-SAA-III-EXT
Record Dates: First submitted 2021-07-12; First posted 2021-07-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Treatment-naive Severe Aplastic Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hetrombopag Olamine (Experimental)
  Interventions: Drug: Hetrombopag Olamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hetrombopag Olamine — Hetrombopag Olamine; once daily
  Arms: Hetrombopag Olamine
Drug: Placebo — Placebo; once daily
  Arms: Placebo

SUMMARY:
This is a multicenter, placebo-control, phase 3 study of hetrombopag in patients with treatment-naive severe aplastic anemia. All subjects who have completed or withdrawn from the HR-TPO-SAA-III study will voluntarily participate in this extension study.

Subjects will receive the same study drug (hetrombopag or placebo) as in study HR-TPO-SAA-III, with the same doses and administration schedule or with modifications based on the actual conditions.

The primary objective of this extension study is to give the subjects participating in the HR-TPO-SAA-III study the continued access to the study drug (hetrombopag or placebo) after the completion of the HR-TPO-SAA-III study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed or withdrawn from the HR-TPO-SAA-III study
2. Subjects who have signed the informed consent form
3. Female and male subjects of childbearing age who agree to take adequate contraceptive measures during the extension study period and within 28 days after the last dose
4. Subjects who have completed the end-of-treatment evaluation in the original study

Exclusion Criteria:

1. Any unstable situation or situation that will compromise the safety of the subject
2. Evidence of clonal cytogenetic abnormalities at the end-of-treatment examination of the HR-TPO-SAA-III study
3. Subjects with uncontrollable hemorrhage and/or infection after standard treatment
4. Subjects who have experienced deep vein thrombosis, myocardial infarction, stroke, or peripheral arterial embolism within 1 year
5. Any situation that may compromise the subject and the safety or compliance thereof during the study

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The ratio of subjects with clonal evolution at 6 months and 18 months | 6 months and 18 months
All SIEs, regardless of whether they are related to the investigational product | 3 years
All SAEs, regardless of whether they are related to the investigational product | 3 years
All AEs resulting in discontinuation and withdrawal from study | 3 years

SECONDARY OUTCOMES:
Red blood cell count | by 1day visit
Hemoglobin | by 1day visit
Platelet count | by 1day visit
White blood cell count | by 1day visit
Neutrophil count | by 1day visit
Reticulocyte count | by 1day visit
The 6-month and 18-month survival rates of subjects | 6 months and 18 months
The recurrence rates at 6 months and 18 months | 6 months and 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China